CLINICAL TRIAL: NCT06295354
Title: Early Variations in Immune Aging
Acronym: EVIA-NL
Status: Terminated | Type: Observational
Why Stopped: Low participant number.
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-17062
Record Dates: First submitted 2024-02-26; First posted 2024-03-06 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2024-10

CONDITIONS: Aging; Aging Well; Immuno Aging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Stool samples
  * Blood samples (isolated cell populations, RNA and DNA)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- 20-30 years old: The target population consists of 1000 participants, equally distributed over different age groups (20-30, 30-40, 40-50, and 50-60 years old) and sex. Main exclusion criteria are any systemic condition or medication apart from cardiometabolic disorders, pregnancy at inclusion or recent vaccinations. Individuals will be compared over time, and age groups will be compared over time and per time point. None of the age groups will get an intervention, the goal is to observationally study them.
  Interventions: Other: No intervention, we just study 'aging'
- 3-40 years old: The target population consists of 1000 participants, equally distributed over different age groups (20-30, 30-40, 40-50, and 50-60 years old) and sex. Main exclusion criteria are any systemic condition or medication apart from cardiometabolic disorders, pregnancy at inclusion or recent vaccinations. Individuals will be compared over time, and age groups will be compared over time and per time point. None of the age groups will get an intervention, the goal is to observationally study them.
  Interventions: Other: No intervention, we just study 'aging'
- 40-50 years old: The target population consists of 1000 participants, equally distributed over different age groups (20-30, 30-40, 40-50, and 50-60 years old) and sex. Main exclusion criteria are any systemic condition or medication apart from cardiometabolic disorders, pregnancy at inclusion or recent vaccinations. Individuals will be compared over time, and age groups will be compared over time and per time point. None of the age groups will get an intervention, the goal is to observationally study them.
  Interventions: Other: No intervention, we just study 'aging'
- 50-60 years old: The target population consists of 1000 participants, equally distributed over different age groups (20-30, 30-40, 40-50, and 50-60 years old) and sex. Main exclusion criteria are any systemic condition or medication apart from cardiometabolic disorders, pregnancy at inclusion or recent vaccinations. Individuals will be compared over time, and age groups will be compared over time and per time point. None of the age groups will get an intervention, the goal is to observationally study them.
  Interventions: Other: No intervention, we just study 'aging'

INTERVENTIONS:
Other: No intervention, we just study 'aging' — No intervention, we just study 'aging'

SUMMARY:
Background:

Despite an increase in lifespan over the last decades, our healthspan lags behind. In our aging population, it is pressing that we prevent age-related morbidities and associated burden on the health care system. Instead of investigating aging in already aged populations, the currently proposed study aims to elucidate the process of immune aging in relation to biological aging, demographic and lifestyle factors in young and midlife adults, and to identify early biomarkers and pathways associated with fast versus slow immune aging and aging endotypes.

Study design:

A single-center, observational prospective cohort study in the Netherlands. Participants from priorly established cohorts will be invited to join the EVIA-study. We will obtain demographic and basic clinical data and biological samples (blood and stool) at baseline and after three years, with a short, yearly online questionnaire in between.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 20 and 60 years;
* Able to communicate orally in Dutch or English;
* Able to give informed consent.

Exclusion Criteria:

* Any systemic disease or condition, or the use of systemic medication, with the exception of the following:

  * Cardiovascular disease and related medication
  * Metabolic syndrome, including diabetes, hypertension, and hyperuricemia
* Pregnancy at inclusion (will be recorded during study);
* Acute illness or fever <1 month before inclusion;
* Received vaccines or antibiotics 3 months before inclusion;
* Participation in an intervention trial;
* Legally incapacitated or unwilling to provide informed consent.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants for each age group will be recruited via invitation. Former participants from the HFGP cohorts will be invited only if they had originally given permission to be approached for future studies. In case insufficient inclusions result from previous cohorts, we will proceed to recruit new healthy volunteers from the Nijmegen region. In that case, we will promote the study via local newspaper(s), social media, and flyers (will be added to the CMO file should this arise). This way, the recruitment is performed as an open invitation, and any willing participants may reach out to the research team via email or telephone.
  This is an observational study to explore natural aging. Participants are not subjected to any intervention.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2024-10-07 (Actual); Primary Completion 2025-01-27 (Actual); Study Completion 2025-03-18 (Actual)

PRIMARY OUTCOMES:
Immunological function | At baseline and after 3 years
  As comprised by cytokine porudction capacity, immunophenotyping, circulating inflammatory markers and metabolomics
Immunological Aging Score | At baseline and after 3 years
  As scored by immune population aging scores, an inflammatory aging score (unpiblished work) and a transcriptomics aging score (idem)
Biological Aging Score | At baseline and after 3 years
  As scored by epigenetic aging (scored by means of DNA methylation), organ aging (Oh et al) and lipidomic aging scores (unpublished)
Metagenomics | At baseline and after 3 years
  From stool microbiome
Genetics and epigenetics | At baseline and after 3 years
  SNPs, telomere attrition, accessible loci
Clinical events | Between baseline and the 3-year timepoint
  Hospital admissions and new medical diagnoses

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud university medical center, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided